CLINICAL TRIAL: NCT00382629
Title: BHT-3009 Immunotherapy in Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayhill Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BHT-3009-03
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple sclerosis; MS; Bayhill; BHT-3009; immunotherapy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — BHT 3009

INTERVENTIONS:
Drug: BHT-3009 0.5 mg
Drug: BHT-3009 1.5 mg
Drug: Placebo

SUMMARY:
The purpose of this study is to determine if BHT-3009 decreases inflammation (measured by gadolinium enhancing MRI lesions) in the brains of people with relapsing remitting multiple sclerosis.

DETAILED DESCRIPTION:
People with multiple sclerosis are thought to have abnormal immunity. Usually the body's immune system attacks only foreign substances, but people with MS have abnormal immunity, where the immune system attacks normal proteins, one of which is a protein found in the brain called MBP (myelin basic protein). This abnormal immunity causes inflammation in the brain resulting in nerve damage. BHT-3009 is a drug that is designed to decrease this abnormal immunity to MBP. BHT-3009 is a DNA plasmid that contains the gene for MBP. Plasmids are circular pieces of DNA that are being tested in clinical trials for their ability to alter patients' immune systems. Two different doses of BHT-3009 will be tested to determine if there are any differences in their safety or effects on inflammation.

Treatment in this study is 3 doses every two weeks for 6 weeks, followed by a dose every 4 weeks for a total of 13 doses in 44 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of multiple sclerosis by the McDonald criteria.
2. Screening cranial MRI demonstrating lesions consistent with MS.
3. One or more relapses within the previous year.
4. Clinically stable (no relapses) for > 50 days before beginning screening procedures and during the screening period.
5. EDSS 0 to 3.5 inclusive.
6. Age > 17 years and < 56 years.
7. Willing and able to give informed consent.
8. WBC >3,000; platelets >100,000; hemoglobin > 10.0 g/dl.
9. AST, ALT, bilirubin < 2.0 x upper limit of normal.
10. Creatinine < 2.0 x upper limit of normal.
11. Negative test for HIV.

Exclusion Criteria:

1. Primary progressive, secondary progressive or progressive relapsing MS.
2. More than 5 gadolinium-enhancing lesions on the first screening MRI.
3. High-dose corticosteroids (e.g. > 500 mg methylprednisolone or equivalent per day for 3 or more days) within 50 days prior to beginning screening procedures.
4. Previous stem cell transplantation, total lymphoid radiation, or cytotoxic therapy.
5. Treatment with interferon, glatiramer acetate or other approved disease-modifying agent for > 180 days (lifetime total of all agents).
6. Treatment with an approved disease modifying agent within 180 days of beginning screening procedures.
7. Previous treatment of MS with an experimental agent including off-label use of approved drugs. (Allowed with approval of the Medical Monitor.)
8. Prior therapy with natalizumab (Tysabri).
9. Pregnant or lactating women.
10. Unwilling to use a medically acceptable form of birth control (e.g. hormonal contraception, intrauterine device, double barriers, sterilization of self or partner).
11. Clinically significant ECG abnormalities (e.g. acute ischemia or life-threatening arrhythmia).
12. Medical condition or social circumstances that would in the opinion of the investigator prevent full participation in the trial or evaluation of study endpoints.
13. Implanted pace makers, defibrillators or other metallic objects on or inside the body that limit performing MRI scans.
14. Known hypersensitivity or allergy to gadolinium.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252
Dates: Start 2006-02; Study Completion 2007-06

PRIMARY OUTCOMES:
Evaluate the effect of BHT-3009 on the mean four-week rate of occurrence of new gadolinium (Gd) enhancing MRI lesions in relapsing remitting MS.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of intramuscular injections of BHT-3009 given for a total of one year.
Evaluate the effect of BHT-3009 on other cranial MRI measures.
Describe the effect of BHT-3009 therapy on relapse rate.
Describe the effect of BHT-3009 on subject disability scores.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Valone, MD, Study Director — Bayhill Therapeutics

REFERENCES:
- See also: Bayhill website — http://www.bayhilltherapeutics.com